CLINICAL TRIAL: NCT01843426
Title: Diagnostic Image Quality and Safety of Low-Volume, Low-Concentration, Iso-Osmolar Contrast Medium in the Computed Tomographic Workup of Patients Considered for TAVR
Brief Title: Aortic Stenosis Pre-Transcatheter Aortic Valve Replacement (TAVR) Procedure CT Scan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro19770
Record Dates: First submitted 2013-04-15; First posted 2013-04-30 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-03

CONDITIONS: Aortic Valve Stenosis
Keywords: Comorbidity
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-volume, Low-concentration contrast (Visipaque 270) CT scan (Experimental): An ECG-synchronized, contrast-medium enhanced CT study of the heart for the evaluation of the aortic root complex and general cardiac morphology will be obtained. This is immediately followed by a CT angiographic study of the chest, abdomen, and pelvis (beyond the femoral heads), which utilizes the same contrast bolus that is injected for evaluating the heart. This latter vascular study serves to evaluate the TAVR deployment catheter access route through the femoral, iliac, and aortic vascular stations. In clinical routine, we have been performing this type of study with total contrast media volumes ranging from 40-120 mL of iodinated contrast material.
  Interventions: Drug: Low-volume, low-concentration contrast (iodixanol - Visipaque 270) CT scan

INTERVENTIONS:
Drug: Low-volume, low-concentration contrast (iodixanol - Visipaque 270) CT scan — An ECG-synchronized, contrast-medium enhanced CT study of the heart for the evaluation of the aortic root complex and general cardiac morphology will be obtained. This is immediately followed by a CT angiographic study of the chest, abdomen, and pelvis (beyond the femoral heads), which utilizes the same contrast bolus that is injected for evaluating the heart. This latter vascular study serves to evaluate the TAVR deployment catheter access route through the femoral, iliac, and aortic vascular stations. In clinical routine, we have been performing this type of study with total contrast media volumes ranging from 40-120 mL of iodinated contrast material.

SUMMARY:
The purpose of this study is to evaluate contrast media volume, safety and 30-day outcome of patients after a computed tomography (CT) scan. The results of this study will help to determine the minimum volume of contrast material that can be used to ensure patient safety while not compromising diagnostic image quality in high-risk patients.

DETAILED DESCRIPTION:
The scholarly rationale for the study is to determine the feasibility of restricting the contrast media volume to 60ml of 270mg Iodine (mgI)/ml iodixanol or less to accomplish sufficient intravascular attenuation for comprehensive CT assessment prior to TAVR. The study will also evaluate the effects of contrast media administration on our subjects' kidney function by performing serum creatinine measurements at baseline, as well as at three days and thirty days after contrast media administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18-90 years of age.
2. Subject must have been referred for a clinically indicated CT prior to TAVR.
3. Subject must provide written informed consent prior to any study-related procedures being performed.
4. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

1. Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:

   * By testing (serum or urine βHCG) within 24 hours before contrast agent administration, or
   * By surgical sterilization, or
   * Post menopausal, with minimum one (1) year history without menses.
2. Subject has an acute psychiatric disorder or is cognitively impaired.
3. Subject is using or is dependent on substances of abuse.
4. Subject is unwilling to comply with the requirements of the protocol.
5. Subject has previously entered this study.
6. Subject has an allergy against iodinated contrast agents.
7. Subject is in acute unstable condition.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Clinically Diagnostic CT Assessments | up to 2 years
  Determine that restricting the contrast media volume to 60ml of 270 mgI/ml iodixanol or less generates clinically diagnostic CT assessments prior to TAVR.

SECONDARY OUTCOMES:
Image Quality | up to 2 years
  Measure contrast media attenuation and determine diagnostic image quality within target structures in the aortic root and the ilio-aortic access route.
Safety | up to 2 years
  Evaluate safety and 30-day outcome of patients regarding survival, renal function, and adverse events (renal failure, dialysis, general morbidity).
Long-term Follow-Up | up to 4 years
  Determine procedural outcome of the TAVR procedure by longer-term patient follow-up after one and two years for device function, position, and paravalvular leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Schoepf, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States